CLINICAL TRIAL: NCT06532344
Title: An Open-label, Uncontrolled Study of ONO-7913 and ONO-4538 in Combination With Modified FOLFIRINOX Therapy, the Standard of Care, as First-line Treatment in Patients With Metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-7913-03
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — magrolimab; Nivolumab; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ONO-7913+ONO-4538+mFFX (Experimental)
  Interventions: Drug: ONO-7913; Drug: ONO-4538; Drug: Oxaliplatin; Drug: Levofolinate; Drug: Irinotecan; Drug: Fluorouracil

INTERVENTIONS:
Drug: ONO-7913 — Specified dose on specified days
  Other Names: Magrolimab
Drug: ONO-4538 — Specified dose on specified days
  Other Names: Nivolumab
Drug: Oxaliplatin — Specified dose on specified days
Drug: Levofolinate — Specified dose on specified days
Drug: Irinotecan — Specified dose on specified days
Drug: Fluorouracil — Specified dose on specified days

SUMMARY:
To investigate the tolerability and safety of ONO-7913 and ONO-4538 used in combination with modified FOLFIRINOX (mFFX therapy), the standard of care, as first-line treatment in patients with metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Untreated metastatic pancreatic cancer
* 2. Life expectancy of at least 3 months
* 3. Patients with ECOG performance status 0 or 1

Exclusion Criteria:

* 1. Patients with severe complication
* 2. Patients with multiple primary cancers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities（DLT） | 28 days
Adverse event(AE) | UP to 30 days after the last dose

SECONDARY OUTCOMES:
Pharmacokinetics（serum concentration of ONO-7913） | Through study completion, an average of 6 months
Pharmacokinetics（serum concentration of ONO-4538） | Through study completion, an average of 6 months
Overall response rate (ORR) | Through study completion, an average of 6 months
Disease control rate (DCR) | Through study completion, an average of 6 months
Overall survival (OS) | Through study completion, an average of 6 months
Progression-free survival (PFS) | Through study completion, an average of 6 months
Duration of response (DOR) | Through study completion, an average of 6 months
Time to response (TTR) | Through study completion, an average of 6 months
Best overall response (BOR) | Through study completion, an average of 6 months
Percentage of change in the sum of tumor diameters of target lesions | Through study completion, an average of 6 months
Maximum percentage of change in the sum of tumor diameters of target lesions | Through study completion, an average of 6 months
Changes in tumor markers (CEA and CA19-9) | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (9):
- Japan (9):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Juntendo University Hospital, Bunkyō-Ku, Tokyo
  - The University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - The Cancer Institute Hospital ofJFCR, Koto-ku, Tokyo
  - Kyorin University Hospital, Mitaka-shi, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - National Cancer Center Hospital, Chūōku

IPD SHARING:
Plan to Share IPD: No